CLINICAL TRIAL: NCT07368530
Title: Radiomics-based Unsupervised Machine Learning Model to Identify Responders to Transarterial Chemoembolization Versus Hepatic Arterial Infusion Chemotherapy in Unresectable Hepatocellular Carcinoma: a Retrospective Cohort Study
Brief Title: Using Machine Learning to Identify Responders to TACE or HAIC for uHCC
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wenzhe Fan, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2026]023
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Hepatocellular Carcinoma (HCC); BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; transarterial chemoembolization; hepatic arterial infusion chemotherapy; machine learning
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE group: Patients with unresectable HCC treated with transarterial chemoembolization
  Interventions: Procedure: Transarterial chemoembolization (TACE)
- HAIC group: Patients with unresectable HCC treated with hepatic arterial infusion chemotherapy
  Interventions: Procedure: hepatic arterial infusion chemotherapy (HAIC)

INTERVENTIONS:
Procedure: Transarterial chemoembolization (TACE) — 1
  Groups: TACE group
Procedure: hepatic arterial infusion chemotherapy (HAIC) — 1
  Groups: HAIC group

SUMMARY:
The goal of this observational study is to learn about the efficacy of Transarterial Chemoembolization (TACE) versus Hepatic Arterial Infusion Chemotherapy (HAIC) in patients with unresectable hepatocellular carcinoma (HCC). The main questions it aims to answer are:

Can distinct imaging phenotype subtypes be identified in unresectable HCC patients using radiomics and unsupervised clustering?

Do these different imaging subtypes show significant differences in treatment efficacy (such as objective response rate, progression-free survival, and overall survival) after receiving TACE or HAIC?

Can this method objectively identify which imaging subtype of patients is more suitable for TACE and which may benefit more from HAIC?

Participants in this study are adult patients diagnosed with unresectable HCC (BCLC stage B or C) who have already undergone complete TACE or HAIC treatment as part of their regular medical care between January 2015 and December 2024. Researchers will retrospectively analyze their existing clinical data and pre-treatment medical images to compare outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with hepatocellular carcinoma (HCC) based on clinical or pathological criteria;
2. Barcelona Clinic Liver Cancer (BCLC) stage B or C, assessed as unresectable by surgical evaluation;
3. Received either TACE or HAIC as the sole interventional treatment modality throughout the treatment course (no crossover between the two modalities allowed);
4. Liver function classified as Child-Pugh Class A or B, or achieved this standard after medical treatment;
5. Performance status (PS) score of 0 or 1.

Exclusion Criteria:

1. Patients with an unclear diagnosis or those with concurrent other malignant tumors;
2. Liver function classified as Child-Pugh Class C or worse, which cannot be improved after hepatoprotective treatment;
3. Patients with severe infections, such as respiratory, biliary tract, or abdominal infections;
4. Patients with severe underlying diseases, particularly immune-related disorders.
5. Patients with severely incomplete or missing baseline or outcome data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable HCC who TACE or HAIC
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of initial treatment until the date of death from any cause, whichever came first, assessed up to 24 months
  Time interval from date of initial treatment until the date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Progression free survival | From date of initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time interval from date of initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Tumor response | From date of initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Defined as the proportion of patients achieving complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) according to mRECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiiated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
This study utilizes existing clinical and imaging data collected as part of routine medical care. The dataset contains detailed and potentially re-identifiable patient information, including medical images, clinical records, and treatment outcomes. Due to institutional data privacy policies, ethical restrictions related to patient confidentiality, and the lack of broad consent from participants for data sharing beyond the scope of this specific research, we are unable to publicly share individual participant data. All data will be stored securely within the hospital's internal research database, and access will be restricted to the study investigators for analysis purposes only. Requests for aggregated or de-identified results may be considered upon reasonable inquiry to the corresponding author, subject to institutional review and compliance with applicable regulations.